CLINICAL TRIAL: NCT02812290
Title: Multi-Centric Observational Study to Analyze the Diagnostic Molecular Features in the Clinical Setting of Lung Allograft Biopsies
Brief Title: Diagnostic and Therapeutic Applications of Microarrays in Lung Transplantation
Acronym: INTERLUNG
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Philip Halloran, Distinguished Professor, University of Alberta
Other Study IDs: ATAGC 03
Record Dates: First submitted 2016-05-31; First posted 2016-06-24 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lung Transplant Rejection
Keywords: antibody mediated rejection; T cell mediated rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lung transplant biopsies taken as per local standard of care.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Lung transplant biopsy bites. — In the second phase of the study, two biopsy bites from the same patient will be collected to assess tissue sampling variability.

SUMMARY:
Objective: To evaluate the potential impact of molecular phenotyping of transbronchial biopsies in lung transplant recipients with allograft dysfunction, and the potential for developing a safer endobronchial mucosal biopsy format.

DETAILED DESCRIPTION:
The current standard for biopsy-based diagnoses of dysfunction of lung transplants is the International Society of Heart and Lung Transplantation (ISHLT) classification applied to transbronchial biopsies, which represents an arbitrary international consensus. Recent data-driven approaches using molecular and conventional technologies indicate that this system produces frequently incorrect diagnoses with potential harm to patients due to inappropriate treatment. especially in relationship to the correct diagnosis of chronic lung allograft dysfunction is a pressing need. To address this unmet need and improve diagnostics in the area of organ transplantation, the Alberta Transplant Applied Genomics Centre (ATAGC, University of Alberta) has developed a new diagnostic system - the Molecular Microscope® Diagnostic System (MMDx) that interprets biopsies in terms of their molecular phenotype. The MMDx, developed first in kidney transplant biopsies with thoroughly established phenotypes, will now be adapted to lung transplant transbronchial biopsies (TBBs). Microarray analysis of lung allograft biopsy specimens will be compared to conventional allograft phenotyping, including clinical, physiologic, radiographic and histological assessment. The present study will use the MMDx™ system to assess and report TBBs, and validate and refine this system in 300 unselected prospectively collected lung TBBs. A subset of the study will examine the third bifurcation mucosal endobronchial biopsies (3BMBs) paired with TBBs from 50 patients to see if the safer 3BMBs can substitute for the TBB to be used by MMDx™. Due to a considerable interest and support from participating Centers, the study is further extended and collected 1032 TBBs and 602 3BMBs from 849 patients. This this is the extension of the INTERLUNG study - INTERLUNGEX.

ELIGIBILITY:
Inclusion Criteria:

* All lung transplant recipients undergoing a biopsy as determined by their surgeon or physician.

Exclusion Criteria:

* Patients who declined participation or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with functioning lung transplant biopsied to determine their graft dysfunction or to confirm good function as per standard of care.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Report the molecular scores (probability) of lung transplant disease in a reference set of 600 transbronchial biopsies. | two years
  Molecular classifier predicts antibody mediated and T cell mediated rejection, and chronic allograft dysfunction.
Report the molecular diagnoses of the MMDx-TBB system | two years
  Compare MMDx readings to standard-of-care TBB histology and clinical diagnosis of CLAD.

SECONDARY OUTCOMES:
Report the molecular scores (probability) of lung transplant disease in a reference set of 600 mucosal endobronchial biopsies. | two years
  Molecular classifier predicts antibody mediated and T cell mediated rejection, and chronic allograft dysfunction.
Report the molecular diagnoses of the MMDx-3BMB system | two years
  Compare MMDx-3BMB readings to MMDx-TBB readings and clinical diagnosis of CLAD
Report the molecular changes over time in medically indicated follow-up biopsies | two years
  Predict and monitor response to anti-rejection treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Halloran, MD, PhD, Principal Investigator — Faculty of Medicine and Dentistry, University of Alberta
Locations (11):
- United States (4):
  - St. Joseph's Hospital and Medical Center 350 West Thomas Road, Floor 8HLT, Phoenix, Arizona
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Division of Pulmonary and Critical Care, Washington University School of Medicine, St Louis, Missouri
  - University of Texas at San Antonio, San Antonio, Texas
- The Alfred Hospital, Monash University, Melbourne, Australia
- Department of Thoracic Surgery, Medical University of Vienna, Vienna, Austria
- Canada (3):
  - Alberta Transplant Applied Genomics Centre, University of Alberta, Edmonton, Alberta
  - Department of Medicine, University of Alberta, Edmonton, Alberta
  - University Health Network, Toronto General Hospital, Toronto, Ontario
- Charles University/Hospital Motol, Prague, Czechia
- Thoracic Surgery Transplant Clinic, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Madill-Thomsen KS, Halloran PF. Precision diagnostics in transplanted organs using microarray-assessed gene expression: concepts and technical methods of the Molecular Microscope(R) Diagnostic System (MMDx). Clin Sci (Lond). 2024 Jun 5;138(11):663-685. doi: 10.1042/CS20220530. PMID 38819301
- [Result] Halloran KM, Parkes MD, Chang J, Timofte IL, Snell GI, Westall GP, Hachem R, Kreisel D, Trulock E, Roux A, Juvet S, Keshavjee S, Jaksch P, Klepetko W, Halloran PF. Molecular assessment of rejection and injury in lung transplant biopsies. J Heart Lung Transplant. 2019 May;38(5):504-513. doi: 10.1016/j.healun.2019.01.1317. Epub 2019 Feb 6. PMID 30773443
- [Result] Halloran K, Parkes MD, Timofte I, Snell G, Westall G, Havlin J, Lischke R, Hachem R, Kreisel D, Levine D, Kubisa B, Piotrowska M, Juvet S, Keshavjee S, Jaksch P, Klepetko W, Hirji A, Weinkauf J, Halloran PF. Molecular T-cell-mediated rejection in transbronchial and mucosal lung transplant biopsies is associated with future risk of graft loss. J Heart Lung Transplant. 2020 Dec;39(12):1327-1337. doi: 10.1016/j.healun.2020.08.013. Epub 2020 Aug 26. PMID 32943286
- [Result] Halloran K, Parkes MD, Timofte IL, Snell GI, Westall GP, Hachem R, Kreisel D, Levine D, Juvet S, Keshavjee S, Jaksch P, Klepetko W, Hirji A, Weinkauf J, Halloran PF. Molecular phenotyping of rejection-related changes in mucosal biopsies from lung transplants. Am J Transplant. 2020 Apr;20(4):954-966. doi: 10.1111/ajt.15685. Epub 2019 Dec 1. PMID 31679176
- [Result] Parkes MD, Halloran K, Hirji A, Pon S, Weinkauf J, Timofte IL, Snell GI, Westall GP, Havlin J, Lischke R, Zajacova A, Hachem R, Kreisel D, Levine D, Kubisa B, Piotrowska M, Juvet S, Keshavjee S, Jaksch P, Klepetko W, Halloran PF. Transcripts associated with chronic lung allograft dysfunction in transbronchial biopsies of lung transplants. Am J Transplant. 2022 Apr;22(4):1054-1072. doi: 10.1111/ajt.16895. Epub 2021 Dec 16. PMID 34850543
- [Result] Halloran K, Mackova M, Parkes MD, Hirji A, Weinkauf J, Timofte IL, Snell GI, Westall GP, Lischke R, Zajacova A, Havlin J, Hachem R, Kreisel D, Levine D, Kubisa B, Piotrowska M, Juvet S, Keshavjee S, Jaksch P, Klepetko W, Halloran PF. The molecular features of chronic lung allograft dysfunction in lung transplant airway mucosa. J Heart Lung Transplant. 2022 Dec;41(12):1689-1699. doi: 10.1016/j.healun.2022.08.014. Epub 2022 Aug 27. PMID 36163162
- [Result] Gauthier PT, Mackova M, Hirji A, Weinkauf J, Timofte IL, Snell GI, Westall GP, Havlin J, Lischke R, Zajacova A, Simonek J, Hachem R, Kreisel D, Levine D, Kubisa B, Piotrowska M, Juvet S, Keshavjee S, Jaksch P, Klepetko W, Halloran K, Halloran PF. Defining a natural killer cell-enriched molecular rejection-like state in lung transplant transbronchial biopsies. Am J Transplant. 2023 Dec;23(12):1922-1938. doi: 10.1016/j.ajt.2023.06.003. Epub 2023 Jun 7. PMID 37295720
- [Result] Mackova M, Gauthier P, Chang J, Hirji A, Weinkauf J, Juvet S, Keshavjee S, Havlin J, Lischke R, Zajacova A, Snell G, Westall G, Halloran PF, Halloran K. Molecular biopsy features associated with baseline lung allograft dysfunction in a multicenter international cohort. J Heart Lung Transplant. 2025 Nov 14:S1053-2498(25)02394-0. doi: 10.1016/j.healun.2025.11.005. Online ahead of print. PMID 41242356
- [Derived] Halloran PF. Integrating molecular and histologic interpretation of transplant biopsies. Clin Transplant. 2021 Apr;35(4):e14244. doi: 10.1111/ctr.14244. Epub 2021 Feb 17. No abstract available. PMID 33595110